CLINICAL TRIAL: NCT00312845
Title: A Randomized, Open-Label, Multicenter Study of VELCADE With Rituximab or Rituximab Alone in Subjects With Relapsed or Refractory, Rituximab Naive or Sensitive Follicular B-cell Non-Hodgkin's Lymphoma
Brief Title: Study of VELCADE and Rituximab in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-LYM-3001
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Bortezomib; Rituximab

ARMS (2):
- Bortezomib + Rituximab (Experimental)
  Interventions: Drug: Bortezomib + Rituximab
- Rituximab (Active Comparator)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Bortezomib + Rituximab — VELCADE for Injection will be administered weekly on Days 1,8,15, and 22 of a 35-day cycle in combination with 4 doses of rituximab once a week on Days 1,8,15, and 22 of Cycle 1 and in combination with a single dose of rituximab on Day 1 of Cycles 2 to 5.
  Arms: Bortezomib + Rituximab
Drug: Rituximab — rituximab once a week on Days 1,8,15, and 22 of Cycle 1, and as a single dose on Day 1 of Cycles 2 to 5 (for a total of 8 doses).
  Arms: Rituximab

SUMMARY:
The purpose of this study is to determine if the combination of VELCADE and rituximab improves progression free survival relative to rituximab alone in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma (B-NHL) who never received rituximab or who have previously responded to rituximab. This is an international study being conducted in the United States and in many countries around the world. A complete list of study locations is listed below.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Man or woman and age 18 years or older
* Diagnosis of follicular B-NHL of the following subtypes (World Health Organization [WHO] classification 1997): follicular lymphoma (FL) (Grades 1 and 2).
* Documented relapse or progression following prior antineoplastic treatment. New lesions or objective evidence of progression of existing lesions must document relapse or progression following the previous therapy.

If any prior regimen included rituximab, the subject must have responded (complete response [CR], unconfirmed complete response [CRu], partial response [PR]), and the time to progression (TTP) from the first dose of rituximab must have been 6 months or more.

* At least 1 measurable tumor mass (greater than 1.5 cm in the longest dimension and greater than 1.0 cm in the short axis) that has not been previously irradiated, or has grown since previous irradiation
* In the opinion of the investigator the decision to initiate treatment is justified to manage the subject's lymphoma
* No active central nervous system lymphoma
* Eastern Cooperative Oncology Group [ECOG] status ≤ 2
* Female subjects must be postmenopausal (for at least 6 months), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at screening.
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* In countries where health authorities have approved the pharmacogenomic testing, subjects or their legally acceptable representatives must have signed a separate informed consent that they agree to participate in the genetic part and protein testing part of the study; participation in the genetic and protein testing component is mandatory for pharmacogenomics testing, but optional for serum protein testing and future testing.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

* Diagnosed or treated for a malignancy other than NHL within 1 year of randomization, or who were previously diagnosed with a malignancy other than NHL and have any radiographic or biochemical marker evidence of malignancy. Subjects with completely resected basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy are not excluded.
* Clinical evidence of a transformation from indolent NHL to a more aggressive form of NHL.
* History of disallowed therapies:

  * Prior treatment with VELCADE
  * Antineoplastic (including unconjugated therapeutic antibodies), experimental, or radiation therapy within 3 weeks before randomization
  * Nitrosoureas within 6 weeks before randomization
  * Radioimmunoconjugates or toxin immunoconjugates within 10 weeks before randomization
  * Stem cell transplant within 6 months before randomization
  * Major surgery within 2 weeks before randomization
* Residual toxic effects of previous therapy or surgery of Grade 3 or worse
* Peripheral neuropathy or neuropathic pain of Grade 2 or worse
* Have received an experimental drug or used an experimental medical device within 21 days before the planned start of treatment.
* History of allergic reaction attributable to compounds containing boron or mannitol
* Known anaphylaxis or immunoglobulin E (IgE)-mediated hypersensitivity to murine proteins or to any component of rituximab including polysorbate 80 and sodium citrate dihydrate
* Concurrent treatment with another investigational agent
* Female subject who is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2006-03; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (206):
- United States (41):
  - East Alabama Medical Center, Opelika, Alabama
  - Central Hematology Oncology Medical Group, Inc, Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - St. Jude Heritage Medical Group, Fullerton, California
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Pacific Shores Medical Group, Long Beach, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - North Valley Hematology Oncology, Mission Hills, California
  - University of California, Irvine Medical Center, Orange, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Norwalk Medical Group, Norwalk, Connecticut
  - Hematology Oncology PC, Stamford, Connecticut
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Innovative Clinical Research of South Florida, Miami, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Emory Univeersity ,Winship Cancer Institute, Atlanta, Georgia
  - Suburban Hematology-Oncology Associates, Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Siouxland Hematolgoy-Oncology Associates, Sioux City, Iowa
  - Kansas City Cancer Center, LLC, Kansas City, Kansas
  - Louisville Oncology, Louisville, Kentucky
  - Hematology & Oncology Specialists, Metairie, Louisiana
  - Sinai Hospital, Baltimore, Maryland
  - Hattiesburg Clinic, Hattesburg, Missouri
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Lancaster Cancer Center, Ltd., Lancaster, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Oncology Consultants, Houston, Texas
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Medical College of Wisconsin Milwaukee, Milwaukee, Wisconsin
- Argentina (3):
  - Higa San Martin, La Plata - Buenos Aires
  - Hospital Professor Rodolfo Rossi, La Plata - Buenos Aires
  - Centro Oncologico Integracion Regional, Mendoza
- Australia (6):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Belgium (11):
  - ULB Erasme, Anderlecht
  - AZ Stuivenberg, Antwerp
  - AZ Sint Jan, Bruges
  - Institute J. Bordet, Brussels
  - Clinique Notre Dame, Charleroi
  - UZ Antwerpen - Universitair Ziekenhuis Antwerpen, Edegem
  - UZ Gent - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Ziekenhuis, Dienst Hematologie, Hasselt
  - CHR La Citadelle, Liège
  - CHU Sart Tilman, Liège
  - Heilig Hart Roeselare, Roeselare
- Brazil (4):
  - Servico de Oncologia do Hospital Sao Lucas da PUC do rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital Brigadeiro, São Paulo
  - Faculdade de Medicina do ABC, São Paulo
- Canada (3):
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Hospital, Toronto, Ontario
  - Juravinski Cancer Centre, Hamilton
- China (9):
  - West China Hospital of Sichuan, Chengdu, Sichuan
  - Cancer Hospital (Institute), CAMS&PUMC, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Affiliated Hospital of the Academy of Military Medical Sciences, Beijing
  - Cancer Center, Sun Yat-Sen University, Guangzhou
  - Peking University Third Hospital, Haidian District Beijing
  - RuiJin Hospital, Shanghai
  - Cancer Hospital - FuDan University, Shanghai
- Bank of Cyprus Oncology Centre, Nicosia, Cyprus
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice, Prague
- Finland (2):
  - Paijat - Hameen Keskussairaala, Lahti
  - Satakunnan Keskussairaala, Pori
- France (7):
  - Institut Bergonie, Bordeaux
  - Clinique Victor Hugo, Le Mans
  - Hopital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Hopital Hotel Dieu, Nantes
  - Service des Maladies due sang - Hopital haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (3):
  - Onkologische Schwerpunktpraxis, Herrsching am Ammersee
  - Universitatsklinikum Munster - Klinik fur Innere Medizin, Münster
  - Praxis für Hämetologie und Oncologie, Würzburg
- Greece (3):
  - Laiko General Hospital of Athens - 1st Internist Clinic - Hematology Department, Athens
  - University General Hospital Attikon - 2nd Department of Internal Medicine - Propedeutic & Research Institute, Athens
  - University Hospital of Patras - Department of Internal Medicine - Hematology Division, Rio Patras
- Hungary (3):
  - Debreceni Egyetem, Orvos- es Egeszsegtudomanyl Centrum, iii. Belgyogyaszati Klinika, Debrecen
  - Petz Aladar County Hospital, Győr
  - SZEgedi Tudomanyegyetem, II Belgyaszati Klinika, Szeged
- India (10):
  - Institution Manipal Hospital, Bangalore
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Apollo Speciality Hospital, Chennai
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - SMS Medical College Hospital, Jaipur
  - Apollo Hospitals, Hyderabad Apollo Hospital Complex, Jubilee Hills
  - Shirdi Saibaba Cancer Hospital, Karnataka
  - Department of Medical Oncology - Regional Cancer Centre, Kerala
  - Regional Cancer Centre, Kerala
  - Tata Memorial Centre, Mumbai
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sorraski Tel Aviv Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Universita degli Studi di Perugia, Perugia
  - Azienda Ospedallera Universitaria Policlinico Tor Vergata, Roma
  - Azienda Sanitaria Ospedaliera Molinette S. Giovanni Battista, Torino
- Mexico (3):
  - Instituto Nacional De Ciencias Medicas Y Nutricion Salvador Zubiran, Delagacion Tlalpan
  - Instituto Nacional De Cancerologia Incan, Delagacion Tlalpan
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez UANL, Monterrey, Nuevo Leon
- Canterbury Health Laboratories, Christchurch, New Zealand
- Poland (9):
  - Klinika Hematologii Instytut Chorob Wewnetrznych, Gdansk
  - Klinika Hematologii CMUJ, Krakow
  - Klinika Hematologii - Uniwersytetu Medycznego, Lodz
  - Klinika Hematologii i Transplantologii Szpiku AM, Lublin
  - Wojskowy Instytut Medyczny - Klinika Hematologii, Warsaw
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Klinika Hematologii AM, Warsaw
  - Klinika Nowotworow Ukladu Chlonnego, Warsaw
  - Katedra i Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku, Wroclaw
- Portugal (4):
  - Servico de Hematologia - Hospital de Dia - Hospital Da Universidade de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, E.P.E. - Departmento de Hematologia, Lisbon
  - Hospital de Dia de Hematologia - Hospital de Santa Maria E.P.E., Lisbon
  - Serviço de Onco-hematologia, Instituto Português de Oncologia do Porto Franscisco Gentil, EPE, Porto
- San Juan VA Medical Center, San Juan, Puerto Rico
- Romania (5):
  - Spitalul clinic de urgenta, Brasov
  - Institutul Clinic Fundeni Clinica de Hematologie, Bucharest
  - Spitalul Universitar de Urgenta Hematologie, Bucharest
  - Spitalul Clinic judetean de urgenta "Sf. Spiridon, Clinica Hematologie, Iași
  - Spitalul Clinic judetean de urgenta Mures, Târgu Mureş
- Russia (22):
  - Arkhangelsk Region Clinical Hospital, Arghangelsk
  - Altay Regional Oncology Dispensary, Barnaul
  - Belgorod Regional Oncology Center, Belgorod
  - Cheliabinsk Regional Oncology Dispensary, Chelyabinsk
  - 1st Republican Clinical Hospital of Udmurtia, Izhevsk
  - Cancer Research Center, Moscow
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Moscow Region Clinical Research Institute, Moscow
  - Semashko Central Clinical Hospital #2, Moscow
  - City Oncology Hospital #62, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Novosibirsk State Medical University, Novosibirsk
  - Medical Scientifical Radiology Center, Obninsk
  - Republikan Hospital named after V.A. Baranov, Petrozavodsk
  - St. Petersburg Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Saint Petersburg Pavlov State Medical University, Saint Petersburg
  - St. Petersburg City Hospital #31, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Tomsk Research Oncology Institute, Tomsk
  - Republican Clinical Hospital of Bashkorkostan, Ufa
  - Ekaterinburg City Clinical Hospital #7, Yekaterinburg
- Slovakia (4):
  - FN F.D. Roosevelt - Oddelenie hematologie, Banska Bysterica
  - Fakultna nemocnica L. Pasteura - Klinika hematologie a onkohematologie, Košice
  - Vychodoslovensky Onkologicky Ustave, a.s., Košice
  - Martinska FN, Klinika hematologie a transfuziologie, Martin
- South Africa (4):
  - GVI Oncology Clinical Trial Unit, Panorama, Cape Town
  - Mary Potter Oncology Centre - Little Company of Mary Hospital, Groenkloof, Pretoria
  - Chris Hani Baragwanath Hospital, Johannesburg
  - East Cape Oncology Centre - St. Georges Hospital, Port Elizabeth
- South Korea (6):
  - Lung Cancer Center - National Cancer Center, Gyeonggi-do
  - Samsung Medical Center - Division of Hematology-Oncology, Department of Medicine, Ilmon-Dong, Kangnam-Ku, Seoul
  - Hematology-Oncology Clinic, Center for Specific Organs Cancer - National Cancer Center, Ilsandong-Gu, Goyang-Si, and Gyeonggi-Do
  - Samsung Medical Center - Department of Internal Medicine, Ilwon Dong, Kangnam-Ku, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Durans I Reynals - Institut Catala d'Oncologia, Barcelona
  - Hospital Germans Trias i Pujol Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- Sweden (3):
  - Onkologiska kliniken Universitetssjukhuset, Lund
  - Centrum for Hematologi Karolinska University Hospital, Stockholm
  - Hematologiska kliniken M54 Karolinska University Hospital, Stockholm
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai
- Ukraine (10):
  - Cherkassy Regional Oncology Dispensary, Cherkassy
  - Dnepropetrovsk Regional Clinical Oncology Dispensary, Dnipro
  - Institute for Emergency and Urgent Medical Assistance named after V.K. Gusak of AMS of Ukraine, Donetsk
  - Khmelnitskiy Regional Hopsital, Khmelnitsky
  - Kiev Center of Marrow Transplantaion, Kiev
  - Krivoy Rog Oncology Dispensary, Kryvyi Rih
  - Institute of Blood Pathology and Transfusional Medicine of AMS of Ukraine, Lviv Clinical Hospital #5, Lviv
  - Ukrainian Medical Stomatological Academy, Poltava Regional Dispensary, Poltava
  - Crimean Republic Clinical Oncology Dispensary, Simferopol
  - Zhitomir Gerbachevsky Regional Clinical Hospital, Zhytomyr
- United Kingdom (6):
  - Aberdeen Royal Infirmary - Department of Haematology, Aberdeen
  - Addenbrooke's Hospital - Department of Haematology, Cambridge
  - University Hospital of Wales, Cardiff
  - Guy's & St. Thomas Hospital, London
  - Derriford Hospital - Department of Haematology, Plymouth
  - Taunton & Somerset Hospital, Taunton

REFERENCES:
- [Derived] Zinzani PL, Khuageva NK, Wang H, Garicochea B, Walewski J, Van Hoof A, Soubeyran P, Caballero D, Buckstein R, Esseltine DL, Theocharous P, Enny C, Zhu E, Elsayed YA, Coiffier B. Bortezomib plus rituximab versus rituximab in patients with high-risk, relapsed, rituximab-naive or rituximab-sensitive follicular lymphoma: subgroup analysis of a randomized phase 3 trial. J Hematol Oncol. 2012 Oct 22;5:67. doi: 10.1186/1756-8722-5-67. PMID 23088650
- [Derived] Coiffier B, Osmanov EA, Hong X, Scheliga A, Mayer J, Offner F, Rule S, Teixeira A, Walewski J, de Vos S, Crump M, Shpilberg O, Esseltine DL, Zhu E, Enny C, Theocharous P, van de Velde H, Elsayed YA, Zinzani PL; LYM-3001 study investigators. Bortezomib plus rituximab versus rituximab alone in patients with relapsed, rituximab-naive or rituximab-sensitive, follicular lymphoma: a randomised phase 3 trial. Lancet Oncol. 2011 Aug;12(8):773-84. doi: 10.1016/S1470-2045(11)70150-4. Epub 2011 Jul 1. PMID 21724462

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib + Rituximab: 1.6 mg/m^2 VELCADE for Injection administered weekly on Days 1, 8, 15, and 22 of a 35-day cycle in combination with 4 doses of 375 mg/m^2 rituximab once weekly on Days 1, 8, 15, and 22 of Cycle 1 and a single dose of 375 mg/m^2 rituximab on Day 1 of Cycles 2 through 5 (for a total of 8 doses of rituximab).
- Rituximab: 375 mg/m^2 rituximab once weekly on Days 1, 8, 15, and 22 of Cycle 1, and as a single dose of 375 mg/m^2 on Day 1 of Cycles 2 through 5 (for a total of 8 doses).
Period: Overall Study
Arm/Group | Bortezomib + Rituximab | Rituximab
Started | 336 | 340
Completed | 237 | 245
Not Completed | 99 | 95
Not completed — Adverse Event | 19 | 5
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 14 | 6
Not completed — Disease Progression | 56 | 77
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib + Rituximab | Rituximab | Total
Number analyzed (Participants) | 336 | 340 | 676
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 243 | 242 | 485
  >=65 years | 93 | 98 | 191
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.12) | 57.3 (12) | 57 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 203 | 367
  Male | 172 | 137 | 309
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
  Portugal | 11 | 12 | 23
  Slovakia | 7 | 8 | 15
  Greece | 1 | 1 | 2
  Thailand | 2 | 1 | 3
  Spain | 9 | 5 | 14
  Ukraine | 13 | 11 | 24
  Israel | 7 | 7 | 14
  Russian Federation | 52 | 55 | 107
  Italy | 14 | 15 | 29
  India | 17 | 24 | 41
  France | 13 | 10 | 23
  Australia | 5 | 3 | 8
  South Africa | 2 | 2 | 4
  China | 46 | 40 | 86
  Korea, Republic of | 4 | 3 | 7
  Finland | 1 | 2 | 3
  United Kingdom | 9 | 10 | 19
  Hungary | 3 | 6 | 9
  Czech Republic | 18 | 17 | 35
  Mexico | 9 | 8 | 17
  Canada | 9 | 10 | 19
  Argentina | 2 | 5 | 7
  Brazil | 18 | 21 | 39
  Belgium | 18 | 19 | 37
  Poland | 24 | 21 | 45
  Romania | 6 | 2 | 8
  Germany | 0 | 3 | 3
  Sweden | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival is defined as time from randomization to progressive disease or death due to any cause, whichever occurs first.
Time Frame: Subjects are followed until progressive disease/death or the end of the study. The median follow up time is 33.9 months.
Population: Intention to treat (ITT) population is defined as all patients randomized to the trial.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bortezomib + Rituximab | Rituximab
Number analyzed (Participants) | 336 | 340
days | 389 [351 to 456] | 334 [278 to 365]
Statistical Analysis 1: Comparison: Bortezomib + Rituximab vs Rituximab; Test type: Superiority or Other; p = 0.039, Log Rank

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as Complete Response (CR) + Complete Response Unconfirmed (CRu) + Partial Response (PR) using International Working Group Criteria (IWGC) and Independent Radiographic Review results and clinical results. The IWGC CR requires complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms, and normalization of lactic dehydrogenase and bone marrow involvement. CRu requires more than 75% reduction in sum of product of nodes (SPD). PR requires moer than 50% reduction in SPD.
Time Frame: Subjects are followed until progressive disease/death or the end of the study. The median follow up time is 33.9 months.
Population: The response-evaluable population was defined as all subjects in the ITT population who received at least 1 dose of VELCADE or rituximab, had at least 1 measurable tumor mass (>1.5 cm in the longest dimension and >1.0 cm in the short axis) at baseline, and had at least 1 post-baseline disease assessment by independent radiology reviewers/IRC.
Measure: Number; unit: participants
Arm/Group | Bortezomib + Rituximab | Rituximab
Number analyzed (Participants) | 315 | 324
participants | 199 | 160
Statistical Analysis 1: Comparison: Bortezomib + Rituximab vs Rituximab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: the end of study
Arm/Group | Bortezomib + Rituximab | Rituximab
Serious Adverse Events (participants affected / at risk) | 59/334 | 37/339
Other Adverse Events (participants affected / at risk) | 288/334 | 232/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Rituximab (N=334) | Rituximab (N=339)
Pneumonia (Infections and infestations) | 7 | 3
Herpes zoster (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Pyrexia (General disorders) | 6 | 2
Asthenia (General disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 4 | 1
Anaphylactic reaction (Immune system disorders) | 2 | 0
Hypotension (Vascular disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Left entricular dysfunction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Meningitis (Infections and infestations) | 0 | 1
Necrotixing fasciitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Rituximab (N=334) | Rituximab (N=339)
Thrombocytopenia (Blood and lymphatic system disorders) | 32 | 13
Chills (General disorders) | 28 | 17
Fatigue (General disorders) | 75 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 46 | 15
Headache (Nervous system disorders) | 42 | 24
Paraesthesia (Nervous system disorders) | 39 | 10
Insomnia (Psychiatric disorders) | 30 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 31
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 15
Rash (Skin and subcutaneous tissue disorders) | 24 | 10
Abdominal pain upper (Gastrointestinal disorders) | 20 | 7
Hepatic function abnormal (Hepatobiliary disorders) | 16 | 11
Nasopharyngitis (Infections and infestations) | 22 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 5
Dizziness (Nervous system disorders) | 20 | 9
Neuralgia (Nervous system disorders) | 23 | 1
Hypertension (Vascular disorders) | 21 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No